CLINICAL TRIAL: NCT01437787
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, 3-Arm Study of SAR302503 in Patients With Intermediate-2 or High-Risk Primary Myelofibrosis, Post-Polycythemia Vera Myelofibrosis, or Post-Essential Thrombocythemia Myelofibrosis With Splenomegaly
Brief Title: Phase III Study of SAR302503 in Intermediate-2 and High Risk Patients With Myelofibrosis
Acronym: JAKARTA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EFC12153; 2011-001897-25 (EudraCT Number); U1111-1121-7170 (Other: UTN)
Record Dates: First submitted 2011-09-16; First posted 2011-09-21 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2015-12

CONDITIONS: Hematopoietic Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — fedratinib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo comparator (Placebo Comparator): once daily X 28 days, orally, empty stomach, approximately same time each day
  Interventions: Drug: Placebo
- SAR302503 400 mg (Experimental): once daily X 28 days, orally, empty stomach, approximately same time each day
  Interventions: Drug: SAR302503
- SAR302503 500 mg (Experimental): once daily X 28 days, orally, empty stomach, approximately same time each day
  Interventions: Drug: SAR302503

INTERVENTIONS:
Drug: SAR302503 — Pharmaceutical form:capsule
  Route of administration: oral
  Arms: SAR302503 400 mg; SAR302503 500 mg
Drug: Placebo — Pharmaceutical form:capsule
  Route of administration: oral
  Arms: Placebo comparator

SUMMARY:
Primary Objective:

* To evaluate the efficacy of daily oral doses of 400 mg or 500 mg of SAR302503 (Investigational Medicinal Product, IMP) compared to placebo in the reduction of spleen volume as determined by magnetic resonance imaging (MRI) (or computed tomography scan in patients with contraindications for MRI).

Secondary Objectives:

* To evaluate the effect on Myelofibrosis (MF)-associated symptoms (key MF symptoms) as measured by the modified Myelofibrosis Symptom Assessment Form (MFSAF) diary.
* To evaluate the Overall Survival of patients treated with either 400 mg/day or 500 mg/day of IMP as compared to placebo.
* To evaluate the Progression Free Survival of patients treated with either 400 mg/day or 500 mg/day of IMP as compared to placebo.
* To evaluate the durability of splenic response.
* To evaluate the safety of IMP.

DETAILED DESCRIPTION:
The expected duration of a patient's treatment in this study is approximately 8 months, based on a maximum 28-day screening period, followed by a ≥6-month (6-cycle) treatment period, and an End Of Treatment (EOT) visit, which should be performed at least 30 days following the last administration of IMP or placebo.

Patients who continue to benefit clinically will be allowed to remain on IMP or placebo beyond the 6-month treatment period until the occurrence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of Primary Myelofibrosis (MF) or Post-Polycythemia Vera MF or Post-Essential Thrombocythemia MF, according to the 2008 World Health Organization and International Working Group of Myelofibrosis Research and Treatment (IWG-MRT) criteria.
* MF classified as high-risk or intermediate-risk level 2, as defined by modified IWG-MRT criteria (IPSS) (according to Cervantes F. et. al.; at screening).
* Enlarged spleen, palpable at least 5 cm below costal margin.
* At least 18 years of age.
* Eastern Cooperative Oncology Group performance status of 0, 1, or 2 at study entry.
* The following laboratory values within 14 days prior to the initiation of IMP or placebo:
* Absolute Neutrophil Count (ANC) ≥1.0 x 10exp9/L
* Platelet count ≥50 x 10exp9/L
* Serum creatinine ≤1.5 x Upper Limit of Normal (ULN)
* Serum amylase and lipase ≤1.5 x ULN

Exclusion criteria:

* Splenectomy.
* Any chemotherapy (eg, hydroxyurea), immunomodulatory drug therapy (eg, thalidomide, interferon-alpha), Anagrelide, immunosuppressive therapy, corticosteroids >10 mg/day prednisone or equivalent, or growth factor treatment (eg, erythropoietin), or hormones (eg, androgens, danazol) within 14 days prior to initiation of IMP or placebo; darbepoetin use within 28 days prior to initiation of IMP or placebo. Patients who have had exposure to hydroxyurea (eg, hydrea) in the past may be enrolled into the study as long as it has not been administered within 14 days prior to initiation of IMP or placebo.
* Major surgery within 28 days or radiation within 6 months prior to initiation of IMP or placebo.
* Prior treatment with a Janus Kinase 2 (JAK2) inhibitor.
* Known active (acute or chronic) Hepatitis A, B, or C; and hepatitis B and C carriers
* AST or ALT ≥2.5 x ULN
* Total Bilirubin:
* Exclude if ≥3.0 x ULN
* Patients with total bilirubin between 1.5-3.0 x ULN must be excluded if the direct bilirubin fraction is ≥25% of the total
* Prior history of chronic liver disease (eg, chronic alcoholic liver disease, autoimmune hepatitis, sclerosing cholangitis, primary biliary cirrhosis, hemachromatosis, non-alcoholic steatohepatitis [NASH])

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2011-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Response Rate (RR), defined as the proportion of patients who have a ≥35% reduction in volume of spleen size at the end of Cycle 6, and confirmed 4 weeks thereafter | 6 months

SECONDARY OUTCOMES:
Symptom Response Rate (SRR): Proportion of patients with ≥50% reduction from baseline to the end of Cycle 6 in the total symptom score. | 6 months
  This assessment will be conducted through the modified MFSAF diary, which will be completed during the week prior to Day 1 of each treatment cycle up to Cycle 6, and during the week prior to the end of Cycle 6.
OS (overall survival) of either 400 mg/day or 500 mg/day of IMP as compared to placebo. | approximately 5 years
PFS (progression free survival) of either 400 mg/day or 500 mg/day of IMP as compared to placebo. | approximately 5 years
Proportion of patients who have ≥25% reduction in volume of spleen size at end of Cycle 6, and confirmed 4 weeks thereafter. | 6 months
Duration of spleen response, measured by MRI (or CT scan in patients with contraindications for MRI. | 2 years
Clinical and laboratory events graded by the NCI CTCAE v4.03. | approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (101):
- United States (9):
  - Investigational Site Number 840014, Scottsdale, Arizona
  - Investigational Site Number 840001, La Jolla, California
  - Investigational Site Number 840012, La Jolla, California
  - Investigational Site Number 840006, Los Angeles, California
  - Investigational Site Number 840013, Baton Rouge, Louisiana
  - Investigational Site Number 840008, Rochester, Minnesota
  - Investigational Site Number 840009, Newark, New Jersey
  - Investigational Site Number 840002, Canton, Ohio
  - Investigational Site Number 840004, Houston, Texas
- Australia (5):
  - Investigational Site Number 036001, Box Hill
  - Investigational Site Number 036005, Herston
  - Investigational Site Number 036003, Randwick
  - Investigational Site Number 036004, Tweed Heads
  - Investigational Site Number 036002, Wodonga
- Investigational Site Number 040001, Vienna, Austria
- Belgium (2):
  - Investigational Site Number 056003, Antwerp
  - Investigational Site Number 056001, Leuven
- Brazil (3):
  - Investigational Site Number 076002, Jaú
  - Investigational Site Number 076004, Porto Alegre
  - Investigational Site Number 076001, Rio de Janeiro
- Canada (3):
  - Investigational Site Number 124001, Montreal
  - Investigational Site Number 124003, Montreal
  - Investigational Site Number 124002, Saint John
- France (7):
  - Investigational Site Number 250006, Marseille
  - Investigational Site Number 250005, Nantes
  - Investigational Site Number 250004, Nîmes
  - Investigational Site Number 250002, Pierre-Bénite
  - Investigational Site Number 250007, Poitiers
  - Investigational Site Number 250003, Toulouse
  - Investigational Site Number 250001, Villejuif
- Germany (4):
  - Investigational Site Number 276006, Aachen
  - Investigational Site Number 276007, Bonn
  - Investigational Site Number 276008, Dresden
  - Investigational Site Number 276001, Mannheim
- Hungary (5):
  - Investigational Site Number 348002, Budapest
  - Investigational Site Number 348001, Debrecen
  - Investigational Site Number 348007, Győr
  - Investigational Site Number 348006, Kecskemét
  - Investigational Site Number 348003, Miskolc
- Ireland (2):
  - Investigational Site Number 372002, Dublin
  - Investigational Site Number 372001, Galway
- Israel (2):
  - Investigational Site Number 376003, Haifa
  - Investigational Site Number 376002, Tel Litwinsky
- Italy (6):
  - Investigational Site Number 380002, Bergamo
  - Investigational Site Number 380007, Bologna
  - Investigational Site Number 380004, Florence
  - Investigational Site Number 380001, Pavia
  - Investigational Site Number 380006, Pavia
  - Investigational Site Number 380003, Varese
- Lithuania (2):
  - Investigational Site Number 440001, Kaunas
  - Investigational Site Number 440002, Klaipėda
- Investigational Site Number 484001, Querétaro, Mexico
- Poland (5):
  - Investigational Site Number 616005, Brzozów
  - Investigational Site Number 616002, Gdansk
  - Investigational Site Number 616006, Lodz
  - Investigational Site Number 616010, Warsaw
  - Investigational Site Number 616003, Wroclaw
- Portugal (4):
  - Investigational Site Number 620005, Coimbra
  - Investigational Site Number 620004, Lisbon
  - Investigational Site Number 620001, Lisbon
  - Investigational Site Number 620003, Porto
- Romania (5):
  - Investigational Site Number 642003, Brasov
  - Investigational Site Number 642004, Bucharest
  - Investigational Site Number 642002, Bucharest
  - Investigational Site Number 642006, Bucharest
  - Investigational Site Number 642001, Timișoara
- Russia (7):
  - Investigational Site Number 643009, Moscow
  - Investigational Site Number 643001, Moscow
  - Investigational Site Number 643010, Nizhny Novgorod
  - Investigational Site Number 643008, Petrozavodsk
  - Investigational Site Number 643005, Saint Petersburg
  - Investigational Site Number 643004, Saint Petersburg
  - Investigational Site Number 643007, Volgograd
- Singapore (2):
  - Investigational Site Number 702002, Singapore
  - Investigational Site Number 702001, Singapore
- South Africa (2):
  - Investigational Site Number 710003, Johannesburg
  - Investigational Site Number 710002, Parktown
- South Korea (7):
  - Investigational Site Number 410002, Bundang-Gu
  - Investigational Site Number 410004, Seoul
  - Investigational Site Number 410003, Seoul
  - Investigational Site Number 410001, Seoul
  - Investigational Site Number 410005, Seoul
  - Investigational Site Number 410006, Seoul
  - Investigational Site Number 410007, Seoul
- Spain (2):
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724002, Madrid
- Sweden (2):
  - Investigational Site Number 752001, Stockholm
  - Investigational Site Number 752002, Uddevalla
- Taiwan (3):
  - Investigational Site Number 158002, Changhua
  - Investigational Site Number 158003, Kaohsiung City
  - Investigational Site Number 158001, Taipei
- United Kingdom (10):
  - Investigational Site Number 826006, Belfast
  - Investigational Site Number 826003, Birmingham
  - Investigational Site Number 826002, Glasgow
  - Investigational Site Number 826004, Leeds
  - Investigational Site Number 826001, London
  - Investigational Site Number 826005, London
  - Investigational Site Number 826007, Manchester
  - Investigational Site Number 826008, Newcastle upon Tyne
  - Investigational Site Number 826009, Oxford
  - Investigational Site Number 826010, Southampton

REFERENCES:
- [Derived] Pardanani A, Harrison C, Cortes JE, Cervantes F, Mesa RA, Milligan D, Masszi T, Mishchenko E, Jourdan E, Vannucchi AM, Drummond MW, Jurgutis M, Kuliczkowski K, Gheorghita E, Passamonti F, Neumann F, Patki A, Gao G, Tefferi A. Safety and Efficacy of Fedratinib in Patients With Primary or Secondary Myelofibrosis: A Randomized Clinical Trial. JAMA Oncol. 2015 Aug;1(5):643-51. doi: 10.1001/jamaoncol.2015.1590. PMID 26181658